CLINICAL TRIAL: NCT04312269
Title: Combining MyoCI With Memory Reactivation to Improve Motor Recovery After Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Marc Slutzky, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP0052149
Record Dates: First submitted 2020-03-09; First posted 2020-03-18 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Stroke
Keywords: Sleep
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcomes assessors and participant are blinded to groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- All phase TMR (Experimental): TMR during every stage of sleep
  Interventions: Other: Targeted Memory Reactivation (TMR)
- Slow-wave sleep (SWS) only TMR (Experimental): TMR during slow-wave sleep only
  Interventions: Other: Targeted Memory Reactivation (TMR)
- Reduced frequency TMR (Experimental): TMR during only subset of sessions
  Interventions: Other: Targeted Memory Reactivation (TMR)
- Sham TMR (Sham Comparator): Patients receive no TMR
  Interventions: Other: Targeted Memory Reactivation (TMR)

INTERVENTIONS:
Other: Targeted Memory Reactivation (TMR) — Targeted memory reactivation (TMR) refers to the process of playing audio cues associated with specific learned material quietly during sleep in order to strengthen consolidation of specific memories during sleep.

SUMMARY:
This study will examine the combination of myoelectric computer interface (MyoCI) training with targeted memory reactivation (TMR) in chronic stroke survivors. The study aims to determine whether this training-plus-sleep combination will generalize to improve arm motor function over an extended training protocol in stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

* Age at enrollment is 21 or older
* Hemiparesis from first ever stroke affecting arm movement at least 6 months prior to screening
* Severe to moderate motor impairment (FMA-UE of 7-40)
* At least some voluntary shoulder and elbow muscle activation

Exclusion Criteria:

* Inability to follow instructions of the MyoCI task
* Visual impairment (such as hemianopia) preventing full view of screen
* Anesthesia or neglect in the affected arm, or visual hemineglect (score of 2 on the NIH Stroke Scale Extinction and Inattention subtest)
* Participation in another study on the affected arm within 6 weeks of enrollment or any pharmacological study
* Inability to understand or follow commands in English due to aphasia or other reason
* Diffuse or multifocal infarcts in both hemispheres
* Substantial arm pain preventing participation for 90 minutes a day
* Spasticity treatment (pharmacological or Botox) within last 3 months
* Ferromagnetic implants that are MRI incompatible

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-02-25 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Wolf Motor Function Test (WMFT) | change from baseline at 6 weeks
  The WMFT evaluates upper extremity function on a continuous scale. It measures the time it takes to perform 15 different tasks, with a time limit of 120 s per task.

SECONDARY OUTCOMES:
Fugl-Meyer Assessment of Upper Extremity (UE) Motor Function | change from baseline at 6 weeks
  The FMA-UE is a measure of impairment. Maximum score is 66 on the motor function portion. Items are scored on a 3-point ordinal scale.
Fugl-Meyer Assessment of Upper Extremity (UE) Motor Function | change from baseline at 10 weeks
  The FMA-UE is a measure of impairment. Maximum score is 66 on the motor function portion. Items are scored on a 3-point ordinal scale.
Motor Activity Log (MAL) | change from baseline at 6 weeks
  The MAL is a validated measure of home-based arm function, both quantity and quality of use in 30 different activities of daily living.
Motor Activity Log (MAL) | change from baseline at 10 weeks
  The MAL is a validated measure of home-based arm function, both quantity and quality of use in 30 different activities of daily living.
Modified Ashworth Scale | change from baseline at 6 weeks
  The Modified Ashworth Scale is a measure of spasticity, which is graded on a scale of 0-4 per joint tested.
Modified Ashworth Scale | change from baseline at 10 weeks
  The Modified Ashworth Scale is a measure of spasticity, which is graded on a scale of 0-4 per joint tested.

CONTACTS AND LOCATIONS:
Overall Officials: Marc W Slutzky, MD/PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Clinical functional outcomes and analyzed EMG (co-activation) will be uploaded and shared upon publication.
Supporting Information: Analytic Code
Time Frame: IPD and associated analytic code will be made available upon publication of research results and will remain available for the duration of the funded project.